CLINICAL TRIAL: NCT00297869
Title: Computer-Assisted Decision Support to Increase the Safety of Prescribing to Older Emergency Department Patients
Brief Title: Using Informatics to Enhance Care of Older Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0311-04B; 2004 Jahnigen Career Award
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Elderly; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): Electronic warnings when providers prescribe a potentially inappropriate medication or an excessively dosed medication (based on estimated creatinine clearance)
  Interventions: Procedure: Computer-Assisted Decision Support

INTERVENTIONS:
Procedure: Computer-Assisted Decision Support — Electronic warnings when providers prescribe a potentially inappropriate medication or an excessively dosed medication (based on estimated creatinine clearance)
  Arms: 2

SUMMARY:
The subjects in this study are physicians working in the Wishard Emergency Department. The purpose of this study is to measure the extent to which information technology (i.e.-computers) improves emergency department care. The objective of our study is to evaluate the use of informatics in the emergency department and specifically to determine if computer reminder systems: 1) reduce the number of unsafe medications prescribed to older adults, 2) assist in more safely dosing of medications to adults of all ages, and 3) increase influenza immunization of eligible older patients in the emergency department.

Interventions: The interventions in this study are computer reminders. When releasing patients from the emergency department, physicians currently write all release orders, including prescriptions, on a computer order entry system that is linked to the Regenstrief Medical Record System. The computerized order entry system will be programmed so that physicians randomized (randomly placed) into the intervention group, the group that will receive the intervention, they will receive one of three types of reminders:

1. The medication prescribed is generally considered unsafe for use in older patients. The reminder will then list appropriate alternatives for this medication.
2. The dose of the prescribed medication is excessive and should be adjusted for the patient's creatinine clearance (or kidney function).
3. This patient may be eligible for influenza vaccination.

The physician will then choose to order or disregard the recommendation. The computer system will automatically record what the physician selected to do. The general outcome of interest is the extent to which the electronic reminders successfully improved physician practice in the emergency department setting. This outcome will be compared to physicians who were randomized to the group that did not receive the reminders (the control group).

ELIGIBILITY:
Inclusion Criteria:

* The subjects of this study will be physician providers and residents and medical students practicing under the supervision of a faculty emergency physician. Specific study subjects will include emergency medicine faculty physicians; emergency medicine and internal medicine residents; emergency medicine, surgery, and internal medicine interns; and medical students taking care of patients in our emergency department.

Exclusion Criteria:

* We will not include the members of the research team in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2005-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Proportion of older ED patients who receive a potentially inappropriate medication | During discharge home from the ED

SECONDARY OUTCOMES:
Proportion of ED patients who receive an excessive dose of a medication that requires dosage adjustment for renal insufficiency | During discharge home from the ED

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M. Terrell, DO, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Wishard Memorial Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Terrell KM, Perkins AJ, Dexter PR, Hui SL, Callahan CM, Miller DK. Computerized decision support to reduce potentially inappropriate prescribing to older emergency department patients: a randomized, controlled trial. J Am Geriatr Soc. 2009 Aug;57(8):1388-94. doi: 10.1111/j.1532-5415.2009.02352.x. Epub 2009 Jun 22. PMID 19549022